CLINICAL TRIAL: NCT00660439
Title: Treatment Effects of Narrative Exposure Therapy on Psychiatric Symptoms and Cortisol Levels in Patients With Posttraumatic Stress Disorder
Brief Title: Treatment Effects of Narrative Exposure Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: PhD Anne Marita Milde, University of Bergen, Department of Biological and Medical Psychology
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NET 40
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treatment group, receives Narrative Exposure Therapy immediately after first assessment. Patients are assessed 1 and 6 months after treatment.
  Interventions: Behavioral: Narrative Exposure Therapy
- B (No Intervention): Waiting list control group, receives no intervention for 3 months after first assessment. A second assessment is then administered and patients receives Narrative Exposure Therapy. Patients are assessed 1 and 6 months after treatment.

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Psychological treatment, with narration of positive and traumatic events in patients history, including "in vivo" exposure of traumatic events. The narrative is written down by the therapist.
  Other Names: NET
  Arms: A

SUMMARY:
This study compares Narrative Exposure Therapy with a Waiting list control group, both consists of traumatized patients with diagnosed Posttraumatic Stress Disorder. The main aim is to investigate if the patients psychiatric symptoms and levels of the stress hormone cortisol will improve more after Narrative Exposure Therapy than the Waiting list (i.e. no intervention).

DETAILED DESCRIPTION:
In this study we want to compare Narrative Exposure Therapy (NET) to Waiting list controls. Adult patients with diagnosed Posttraumatic Stress Disorder following different types of trauma, will be included. Clinicians in psychiatric outpatient clinics will treat patients with NET, either immediately after assessment, or after a second assessment 3 months later. All patients will also be assessed 1 and 6 months after treatment completion. All patients will be assessed for psychiatric symptoms by the Mini International Neuropsychiatric Interview (version 5.0.0) and the Clinician-Administered PTSD Scale. Patients will also answer several questionnaires (IES-R, SCL-90, BDI-II, DES and UCL). Baseline level of the stress hormone cortisol will be collected in saliva for measuring the diurnal cycle. We will investigate if patients with Posttraumatic Stress Disorder will show more symptom improvement with NET than those on the waiting list (i.e. no intervention) in addition to measuring potential differences in cortisol between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Posttraumatic Stress Disorder (PTSD)
* Age above 18 years
* Understands, speaks and writes Norwegian
* Informed, written consent

Exclusion Criteria:

* Active psychosis
* Active suicidality
* Serious self mutilation
* Active alcohol or drug abuse
* Serious dissociative symptoms
* Disease in nervous system or head injury
* Hormonal disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Psychiatric symptoms | 1 and 6 months after treatment

SECONDARY OUTCOMES:
Cortisol in saliva | 1 and 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marita Milde, PhD, Study Director — University of Bergen
Locations (1):
- Western Norway Violence and Traumatic Stress Resource Centre, Bergen, Norway